CLINICAL TRIAL: NCT02667977
Title: Reexamining Hypotonic Intravenous Fluid Use in Pediatric Patients With Gastroenteritis.
Brief Title: Reexamining Hypotonic Intravenous Fluid Use
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty getting labs in this setting. After pilot study, this study was not continued.
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Principal Investigator, Waheeda Samady, MD, Pediatric Hospitalist, Ann & Robert H Lurie Children's Hospital of Chicago
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: 2014-15901
Record Dates: First submitted 2014-10-13; First posted 2016-01-29 (Estimated); Last update posted 2016-01-29 (Estimated); Status verified 2016-01

CONDITIONS: Hyponatremia
Keywords: fluids, pediatric, gastroenteritis
MeSH Terms: conditions — Hyponatremia; Gastroenteritis | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Active Comparator): These patients will receive Dextrose 5% and 0.9 NS in their maintenance IV fluids
  Interventions: Other: 0.9 Normal Saline
- Group 2 (Active Comparator): These patients will receive Dextrose 5% and 0.45 NS in their maintenance IV fluids
  Interventions: Other: 0.45 Normal Saline

INTERVENTIONS:
Other: 0.9 Normal Saline — Use of 0.9 Normal Saline for maintenance IV fluids
  Arms: Group 1
Other: 0.45 Normal Saline — Use of 0.45 Normal Saline for maintenance IV fluids
  Arms: Group 2

SUMMARY:
The study aim is to isolate a single type of patient (pediatric patient with acute gastrointestinal symptoms) and evaluate the use of hypotonic (0.45 NS) vs. isotonic (0.9 NS) fluids in these patients in regards to changes in their serum sodium and iatrogenic hyponatremia.

DETAILED DESCRIPTION:
This study will be a randomized patient-blinded 0.45 NS-controlled clinical trial evaluating children ages 6 months to 16 years presenting to the Emergency Department (ED) at Ann & Robert H. Lurie Children's Hospital of Chicago (Lurie Children's) with vomiting and/or diarrhea requiring intravenous fluid therapy. Children will be treated with fluid boluses per ED physician's discretion as is standard of care. After this initial intravenous therapy, children will be admitted to the medical observation unit or general medicine floor for additional fluid therapy. Per standard of care, they will be evaluated clinically by the treating physician who will determine if any additional 0.9 NS boluses are required and administer them at that time. Per standard of care, the treating physician will obtain the information needed to complete the admission history and physical documentation and based on this information will be able to determine if the patient is eligible for the study. The treating physician will complete the Initial Screening Form to document whether the patient is eligible. If a patient is eligible, the treating physician will obtain consent or inform investigators of the patient so that they may obtain consent (depending on whether the treating hospitalist has been trained to obtain consent). For patients who consent to participate, information from the admission History and Physical exam will be extracted on Study Form A. Recruitment will occur only at Lurie Children's. The consent form will provide written information for the family; there are no other recruitment materials. A sign with a reminder about the study will be posted in physician areas.

Those who are eligible and consent to participate in the study will be randomized to receive either 5% dextrose containing 0.45 NS or 5% dextrose with 0.9 NS for their maintenance fluids (see table below). If the treating physician would like to include potassium in the IVF, the potassium concentration will be the standard potassium concentration in both groups (20 mEq/liter). The use of potassium at this concentration is part of standard of care unless patients have a contraindication to its inclusion; this decision made by the treating physician will not alter inclusion in the study and the use of potassium will not impact the results. Block randomization will be utilized using sequential envelopes which will contain the preselected fluid type. This sealed envelope will be opened by the attending hospitalist who will put in the fluid orders. Fluids will be covered by opaque bags so that patients and parents will be blinded to study fluid type. Attending hospitalist physicians and nursing staff will not be blinded to study fluids as all data for this study are objective measurements and our primary outcome is an objective laboratory measurement. The standard fluid administration rate determined by patient weight will be used and this same formula will be applied for both groups. Baseline electrolytes and blood pressure will be checked upon acceptance in the study (prior to maintenance fluid administration) and at 8 hours. Patients in the study will have a basic electrolyte panel drawn through their IV catheter at the beginning of the study prior to the start of their IVF. We will follow standardized protocol for obtaining labs from the IV catheter. If sample cannot be obtained this way, we will obtain them through via a blood draw from the vein if the family agrees. These laboratory studies will be ordered by the physician and completed by trained nursing and/or laboratory staff. This study requires 0.5ml of blood and will provide baseline blood levels of sodium, chloride, bicarbonate, potassium, and glucose. Complete medical and family historical data and socio-demographic information is obtained on all patients as part of the routine admission to the hospital and this information will be extracted from the patient chart for comparison of the two groups.

A majority of patients who are admitted for IVF are either unable to take fluids by mouth or take insufficient amounts of fluids, especially during their first 8 hours of their hospitalization. We anticipate most patients being NPO (nothing by mouth) or on clear fluid diets in the first 8 hours of the hospital stay, reducing oral salt intake. Information regarding oral fluid intake during the first 8 hours will also be extracted from patient chart (intake and output charting). Patients will be otherwise treated per the discretion of their physician for all other aspects of their care, including decision to stop maintenance IVF therapy. After 8 hours, the study IVF will be removed and a second basic electrolyte panel will be obtained. This will provide information about the change in blood sodium levels as well as other electrolytes. After study fluids have been removed and blood samples have been obtained, the treating physician may choose to continue IVF with either type of fluid or discontinue fluids. If the patient does not require IVF for the full 8 hours, the second blood sample will be obtained only if the patient was on the study IVF for >5 hours. In this circumstance, the second blood draw will be obtained whenever the treating physician decides to stop the study IVF. If the IVF are stopped earlier than 5 hours, the primary outcome of a change in sodium of >3 is less relevant. Thus, the patient will be removed from the study and a second blood sample will not be obtained.

This study will be conducted entirely during the hospitalization period. Based on a preliminary study we conducted evaluating 103 patients admitted with nausea, diarrhea, and dehydration, the average length of stay for intravenous fluids was 63 hours with greater than 99% of patients needing more than 8 hours of intravenous fluids. Thus, this study would be conducted within the first 8 hours of therapy and will not extend either length of stay or IVF administration. No additional clinic visitations, hospitalizations, or outpatient resources will be utilized. This study will involve laboratory studies but does not involve radiographic studies or other invasive procedures.

ELIGIBILITY:
Inclusion Criteria:

* Children 6 months to 16 years of age
* Symptoms of acute gastroenteritis (acute vomiting and/or diarrhea; symptoms of the "stomach flu")
* Admission to the hospital
* Requiring maintenance IVF as determined by the inpatient attending clinical judgment.

Exclusion Criteria:

* Age <6 months or age >16 years
* Weight >60 kg
* Admission to the PICU
* Chronic kidney disease
* Endocrine disorders
* Liver or heart disease
* Malignancies
* Human immunodeficiency virus
* Cystic fibrosis
* Epilepsy
* Guillan Barre Syndrome
* Multiple sclerosis.
* Any diuretic medications or medication known to affect ADH secretion
* Abnormal baseline sodium concentration (<133 mEq/L or > 147 mEq/L)
* Abnormal baseline systolic blood pressure (>95% based on age and height normative values)
* Hypotonic or isotonic fluids is deemed contraindicated
* Receives any additional intravenous fluids (NS or lactated ringer boluses) after study fluids have been initiated
* Taking a full diet at the time of admission
* Parents or legal guardians cannot be reached for consent
* Parents and children do not speak English or Spanish as their primary language
* High volume diarrhea (>3 loose stools per day) for a >1 week duration

Ages: 6 Months to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2014-10; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Change in sodium | 8 hours

CONTACTS AND LOCATIONS:
Overall Officials: Waheeda Samady, MD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Ann and Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois, United States